CLINICAL TRIAL: NCT04402359
Title: Comparative Study Between Usage of Meropenem/Gentamicin Versus Ceftazidime/Avibactam in the Treatment of ARDS Induced by Both Lung Trauma and VAP
Brief Title: Usage of Meropenem/Gentamicin Versus Ceftazidime/Avibactam in ARDS
Status: Completed | Type: Observational
Sponsor: King Abdul Aziz Specialist Hospital (Network)
Responsible Party: Sponsor
Other Study IDs: ICU-3-20
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Meropenem; avibactam, ceftazidime drug combination; Ventilators, Mechanical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Group A: Patients of Group A received meropenem one gram slowly IV infusion every 8 hours for 14 days and gentamicin 7 milligram (mg)/ Kilogram body weight per day slowly IV infusion once daily only for one week after ventilator for 2 weeks
  Interventions: Drug: meropenem; Device: ventilator
- Group B: received ceftazidime 2 grams and avibactam 500 mg every 8 hours for 14 days in solution for injection(sodium chloride 9 mg/mL (0.9%), sodium chloride 4.5 mg/mL, dextrose 25 mg/mL, 0.45% sodium chloride, 2.5% dextrose and/or Lactated Ringer's solution). The solution for injection should be administered over 120 minutes.after ventilator for 2 weeks
  Interventions: Drug: ceftazidime 2 grams and avibactam 500; Device: ventilator

INTERVENTIONS:
Drug: meropenem — meropenem one gram slowly IV infusion every 8 hours for 14 days
  Groups: Group A
Drug: ceftazidime 2 grams and avibactam 500 — received ceftazidime 2 grams and avibactam 500 mg every 8 hours for 14 days in solution for injection(sodium chloride 9 mg/mL (0.9%), sodium chloride 4.5 mg/mL, dextrose 25 mg/mL, 0.45% sodium chloride, 2.5% dextrose and/or Lactated Ringer's solution).
  Other Names: Avycaz
  Groups: Group B
Device: ventilator — all patients selected to be ventilated for 14 days

SUMMARY:
This was a prospective double blind study conducted on 200 polytrauma patients admitted to King Abdul-Aziz Specialized Hospital, Taif, KSA between July 2018 and December 2019 in surgical ICU. All patients were having severe chest trauma, contused lungs either with or without severe head trauma.

DETAILED DESCRIPTION:
Patients of Group A received meropenem one gram slowly IV infusion every 8 hours for 14 days and gentamicin 7 milligram (mg)/ Kilogram body weight per day slowly IV infusion once daily only for one week, while patients of Group B received ceftazidime 2 grams and avibactam 500 mg every 8 hours for 14 days in solution for injection(sodium chloride 9 mg/mL (0.9%), sodium chloride 4.5 mg/mL, dextrose 25 mg/mL, 0.45% sodium chloride, 2.5% dextrose and/or Lactated Ringer's solution). The solution for injection should be administered over 120 minutes. • Temperature was measured every 3 hours for 2 weeks. • ABG was done every 8 hours for 2 weeks. • CBC including white cell count was done daily and for 2 weeks. • Complete renal functions daily (urea and creatinine serum level) for 2 weeks. Any patient showing rise in the creatinine level was recorded and excluded from the study. • Chest X-ray for all the patients was ordered after intubation and with onset of ventilation and every 24 hours for 2 weeks. • All patients received anti-stress (Omeprazole 20 mg IV every 12 hours). • Oro-gastric tubes were inserted to all patients and feeding was started within 24 hours.Daily evaluation for conscious level and need for sedation and ventilation were done for all patients. • Tracheobronchial lavage was obtained by bronchoscopy 2 times a week and sent for qualitative culture for 2 weeks. • Blood culture was also taken 2 times per week for 2 weeks. • The planned duration of the study is two weeks from diagnosis of VAP and starting the antibiotics so any patients who failed to be weaned within this period were considered morbidity and recorded.

ELIGIBILITY:
Inclusion Criteria

patients with respiratory failure diagnosed by ABG,chest Xray, and clinical by Arterial oxygen low saturation.

Exclusion Criteria:

* Any other types of respiratory failure rather than trauma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 polytrauma patients admitted to King Abdul-Aziz Specialized Hospital, Taif, KSA between July 2018 and December 2019 in surgical ICU.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2019-12-28 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
systemic change of tissue oxygenation | 2 weeks
  improvement of arterial partial pressure of oxygen

CONTACTS AND LOCATIONS:
Locations (1):
- King abd el Aziz specialist hospital, Ta'if, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
To evaluate and compare the effect of use of combination of meropenem/gentamicin versus the use of ceftazidime/avibactam in the treatment of ARDS induced by both VAP and lung contusion and early weaning from the ventilator and compare their effect on the mortality rate.